CLINICAL TRIAL: NCT07359300
Title: A Randomized Controlled Clinical Trial Comparing Cyanoacrylate and Sutures for Free Gingival Graft Stabilization
Brief Title: Cyanoacrylate Versus Sutures for Free Gingival Graft Stabilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Kübra Burcu Yıldırım, PhD, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YEDITEPE-FGG-2019-01
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Insufficient Keratinized Tissue; Gingival Recession; Mucogingival Defects
Keywords: Free gingival graft; Cyanoacrylate; Sutures; Keratinized tissue; Randomized clinical trial
MeSH Terms: conditions — Gingival Recession | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups to receive free gingival graft stabilization using either butyl-cyanoacrylate tissue adhesive or conventional sutures.
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome measurements were performed by an examiner blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyanoacrylate Stabilization Group (Experimental): Free gingival grafts were stabilized using butyl-cyanoacrylate tissue adhesive following standard free gingival graft surgery.
  Interventions: Procedure: Free Gingival Graft Stabilization With Butyl-Cyanoacrylate
- Suture Stabilization Group (Active Comparator): Free gingival grafts were stabilized using non-resorbable polypropylene sutures following standard free gingival graft surgery.
  Interventions: Procedure: Free Gingival Graft Stabilization With Sutures

INTERVENTIONS:
Procedure: Free Gingival Graft Stabilization With Butyl-Cyanoacrylate — Stabilization of free gingival grafts using butyl-cyanoacrylate tissue adhesive following standard free gingival graft surgery.
  Arms: Cyanoacrylate Stabilization Group
Procedure: Free Gingival Graft Stabilization With Sutures — Stabilization of free gingival grafts using non-resorbable polypropylene sutures following standard free gingival graft surgery.
  Arms: Suture Stabilization Group

SUMMARY:
This randomized controlled clinical trial evaluated the effectiveness of butyl-cyanoacrylate tissue adhesive compared with conventional sutures for stabilization of free gingival grafts. Twenty-four patients with insufficient keratinized tissue were randomly assigned to either cyanoacrylate or suture stabilization following free gingival graft surgery. Clinical parameters, graft dimensional changes, patient-reported postoperative discomfort, and operative time were assessed over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Presence of ≤1 mm of keratinized tissue and/or Miller Class I gingival recession ≤2 mm affecting one to four mandibular anterior teeth
* Vital teeth in the surgical area
* Good oral hygiene following initial periodontal therapy (full-mouth plaque score and full-mouth bleeding score ≤20%)
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

* Current smokers
* Pregnancy or lactation
* Use of systemic antibiotics within the previous 6 months
* History of periodontal surgery in the study area
* Ongoing orthodontic treatment
* Systemic conditions that could affect periodontal healing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Keratinized Tissue Width | Baseline and 6 months postoperatively
  Change in keratinized tissue width measured at the surgical sites using a periodontal probe.

SECONDARY OUTCOMES:
Total Graft Surface Area (TGSA) | Baseline, 1 month, 3 months, and 6 months postoperatively
  Changes in total graft surface area assessed using standardized clinical photographs and digital measurements.
Vertical Graft Height (VGH) | Baseline, 1 month, 3 months, and 6 months postoperatively
  Changes in vertical graft height assessed using standardized clinical photographs and digital measurements.
Probing Depth (PD) | Baseline and 6 months postoperatively
  Changes in probing depth measured at the surgical sites using a periodontal probe.
Vertical Recession (VR) | Baseline and 6 months postoperatively
  Changes in vertical gingival recession measured at the surgical sites using a periodontal probe.
Full-Mouth Plaque Score (FMPS) | Baseline and 6 months postoperatively
  Changes in full-mouth plaque score assessed to evaluate oral hygiene status.
Full-Mouth Bleeding Score (FMBS) | Baseline and 6 months postoperatively
  Changes in full-mouth bleeding score assessed to evaluate periodontal inflammation.
Postoperative Pain and Discomfort | Day 0 to Day 6 postoperatively
  Patient-reported postoperative pain and discomfort assessed using a visual analogue scale (VAS).
Operative Time | During the surgical procedure
  Duration of the surgical procedure measured from the initial incision to completion of graft stabilization.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No